CLINICAL TRIAL: NCT03253536
Title: Prospective Observational Trial to Evaluate Quality of Life After Stereotactic Ablative Radiation Therapy in Patients With Hepatocellular Carcinoma
Acronym: LIVERCARE
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Falk Roeder, Consultant Radiation Oncology, Ludwig-Maximilians - University of Munich
Other Study IDs: Livercare
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Cancer; Quality of Life; Stereotactic Body Radiation Therapy; Observational
Keywords: Hepatocellular Cancer; Quality of Life; stereotactic body radiation therapy; observational
MeSH Terms: conditions — Liver Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- entire cohort: none (observational study)
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — none (observational study)

SUMMARY:
Prospective single arm, single center observational study to evaluate Quality of Life (Qol) after stereotactic body radiotherapy for patients with hepatocellular cancer. Patients will receive work-up, treatment and follow-up exclusively as routinely done except additional quality of life measurements. Qol will be measured by standardized and validated EORTC questionaires at different time points during routine follow-up.

DETAILED DESCRIPTION:
Prospective single arm, single center observational study to evaluate Quality of Life (Qol) after stereotactic body radiotherapy (SBRT) for patients with hepatocellular cancer (HCC). Patients will receive work-up, treatment and follow-up exclusively as routinely done except additional quality of life measurements. This will include contrast-enhanced liver MRI or CT and placement of fiducials if necessary. Radiation treatment planning will be based on contrast-enhanced fourdimensional computed tomography (4D-CT) with abdominal compression. Target volume definition will use an internal target volume (ITV) concept. Dose prescription and fractionation will be prescribed individually based on lesion size, localisation, movement and liver function according to institutional standards. Qol will be measured by standardized and validated EORTC questionaires (QLQ C-30 and HCC 18) at baseline, at the end of SBRT, during follow up at 6 weeks, 3,6,12,24,36,48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* histologically or radiologically proven hepatocellular carcinoma
* 1-3 lesions suitable for stereotactic radiation therapy
* indication for SBRT according to multidisciplinary board evaluation
* age >= 18 years
* written informed consent for study participation
* mental and verbal ability to complete standardized questionaires according to assessment by investigator (physician)

Exclusion Criteria:

* age < 18 years
* prior HCC specific systemic therapy
* concurrent oncological systemic treatment
* distant metastases
* inadequate ability tobe compliant with the protocol or to complete standardizes questionaires
* inability to receive contrast-enhanced planning CT
* missing ability to give informed consent
* legal custody

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients receiving routine SBRT to 1-3 intrahepatic HCC lesions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2022-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 60 months
  Quality of life

SECONDARY OUTCOMES:
acute toxicity | 3 months
  physician-related acute toxicity
late toxicity | 6, 12, 24, 36, 48, 60 months
  physician-related late toxicity
response | 3 months
  response to treatment according to imaging
local control | 60 months
  absence of regrowth inside the treated lesion
hepatic control | 60 months
  absence of regrowth or onset of new lesions inside the liver
distant control | 60 months
  absence of extrahepatic progression
freedom from treatment failure | 60 months
  absence of disease progression other than death
overall survival | 60 months
  absence of death of any cause
pattern of recurrence | 60 months
  pattern of recurrence
correlation Qol with acute toxicity | 3 months
  correlation Qol with acute toxicity
correlation Qol with late toxicity | 6, 12, 24, 36, 48, 60 months
  correlation Qol with late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Falk Roeder, MD, Principal Investigator — Department of Radiation Oncology, University Hospital, LMU Munich
Locations (1):
- Department of Radiation Oncology, University Hospital, LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No